CLINICAL TRIAL: NCT00295217
Title: MR Guided Focused Ultrasound Surgery in the Treatment of Uterine Fibroids: Clinical Study to Validate the Changes to ExAblate 2000 Device
Brief Title: MR Guided Focused Ultrasound Surgery in the Treatment of Uterine Fibroids: Software V4.2 Validation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InSightec (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF017; Continued Access
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Uterine Fibroids; Uterine Leiomyomas
Keywords: Fibroids; Uterine Leiomyomas; ExAblate; MrgFUS
MeSH Terms: conditions — Leiomyoma; Myofibroma

INTERVENTIONS:
Device: ExAblate 2000

SUMMARY:
The goal of this study is to validate the new ExAblate Application software V4.2 by developing additional data that shows the safety of this treatment. The ExAblate is intended to ablate uterine fibroid tissue in pre- or peri-menopausal women with symptomatic uterine fibroids who desire a uterine sparing procedure. Patients must have a uterine size of less than 24 weeks and not seeking treatment for reasons of improving fertility.

ELIGIBILITY:
Inclusion Criteria:

1. Women who present with symptomatic uterine fibroids and are not seeking treatment for the reason of improving fertility.
2. Able and willing to give consent and able to attend all study visits.
3. Patient is pre or peri-menopausal (within 12 months of last menstrual period).
4. Able to communicate sensations during the ExAblate procedure.
5. Uterine fibroids, which are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
6. Fibroids(s) clearly visible on non-contrast MRI.

Exclusion Criteria:

1. Metallic implants that are incompatible with MRI
2. Sensitive to MRI contrast agents
3. Severe claustrophobia that would prevent completion of procedure in MR unit
4. Who are pregnant or desire to become pregnant in the future. Pregnancies following ExAblate treatment could be dangerous for both mother and fetus.
5. Pedunculated fibroids
6. Active pelvic inflammatory disease (PID)
7. Active local or systemic infection
8. Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia
9. Intrauterine device (IUD) anywhere in the treatment path
10. Dermoid cyst of the ovary anywhere in the treatment path
11. Extensive abdominal scarring that cannot be avoided by redirection of the beam (e.g., due to Caesarean section or repeated abdominal surgeries)
12. Undiagnosed vaginal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
In this IDE for the 4.2 ExAblate system, the goal is evaluation of the new features to confirm that they do not introduce any new safety issues.

CONTACTS AND LOCATIONS:
Overall Officials: George Holland, M.D., Principal Investigator — Lahey Clinic; Mark Shaman, M.D., Principal Investigator — KNI; Robert Min, M.D., Principal Investigator — Cornell; Anne Roberts, M.D., Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - University of California at San Diego, La Jolla, California
  - Lahey Clinic, Burlington, Massachusetts
  - KNI, Kalamazoo, Michigan
  - Cornell Vascular, New York, New York

REFERENCES:
- See also: Sponsor web page — http://www.insightec.com